CLINICAL TRIAL: NCT04950062
Title: Effect of High Intensity Interval Training Versus Intermittent Fasting 16/8 Protocol on Functional Capacity Among Overweight Subjects
Brief Title: High Intensity Interval Training Versus Intermittent Fasting on Functional Capacity Among Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Manar Elbaz, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Manar_MSc
Record Dates: First submitted 2021-06-12; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): Group A included 30 subjects who will participate in high intensity interval training on a treadmill for 12 weeks, 3 times/week.
  Interventions: Other: High Intensity Interval Training
- Intermittent fasting (Active Comparator): Group B that included 30 subjects will participate in intermittent fasting for 12 weeks, 3 times/week.
  Interventions: Other: Intermittent Fasting 16/8 Protocol

INTERVENTIONS:
Other: High Intensity Interval Training — 1. Warming up period for 5 min at an intensity corresponding to 65-75% of heart rate maximum (HRmax).
  2. Training phase for 30 min divided into four sets of 4-min length each at intensity equals 80-90% of HRmax interspersed by 3 minutes low intensity walking at the level of 65-75% of HRmax.
  3. Cooling down period for 5 min of at 50-60% of the HRmax. All subjects will be trained at the lower intensity limit for the first 2 weeks of the program before increasing the intensity levels toward the upper limit.
  Arms: High intensity interval training
Other: Intermittent Fasting 16/8 Protocol — Every subject will be instructed to fast a fixed 16 hours followed by 8 hours of eating every day through the whole study period based on their life and sleeping style. During fasting, zero-calorie coffee, tea and water intake will be permitted. Beverages containing calories were consumed during the feeding hours each day. All subjects will be instructed about their optimum caloric requirement based on their basal metabolic rate that will be calculated in advance to avoid over consumption of food on severe caloric restriction as we like to investigate the effect of this way of fasting on reducing weight and improving functional capacity.
  Arms: Intermittent fasting

SUMMARY:
The purpose of the study is to compare the effect of high-intensity interval training and intermittent fasting on improving body weight and functional capacity among overweight subjects.

DETAILED DESCRIPTION:
Exercise improves cardiorespiratory fitness, muscle strength, endurance, body composition, and decreases visceral fat. The, increase in physical activity and modification of eating behaviors are the first line of interventions given because of their low costs and low risks of complications.

Most commonly, the continuous exercise of moderate intensity, that has to be performed several days of the week to get target benefits have been used, on the other hand, different forms of training which aim to reduce time spent exercising by increasing exercise intensity have been considered as an alternative to increasing adherence to the training program which is supported by some researches that may have greater benefits as high intensity interval training improves the vascular function of the muscle capillary density and endothelial nitric oxide synthase(eNOS) levels. But there are some overweight people even some of the young people have restriction to perform exercise programs due to any medical problem that could interfere with exercise.

So, searching for optimal dietary interventions for obesity is still ongoing, but the modification in eating behaviors are hampered by difficulties in coping with a different diet. So, the diet with a fasting component that will be used in this study may be more effective than other complex and restrictive diets as it essentially limits the caloric intake to a specified period without major diet composition changes.

So, the aim of this study is to compare the effect of high-intensity interval training and intermittent fasting on improving body weight and functional capacity among overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to meet all the following criteria in order to participate in the study:

  1. Overweight subjects with age from 25 to 35 years.
  2. Body mass index will be range from 25 to 29.9 kg/m2.
  3. Waist circumference ≥ 80 cm2.
  4. A minimum of 70% of exercise program and diet regimen compliance will be required in order to be included.

Exclusion Criteria:

* Subjects with the following disorders will be excluded from participating in this study:

  1. Musculoskeletal, cardiovascular disorders.
  2. Asthma, chronic obstructive pulmonary diseases.
  3. Any systemic disease or condition that might reduce adherence or tolerance to exercise or fasting.
  4. History of stroke.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Assessing the change in Vo2max | Baseline and 2 months post-intervention
  Assessment via using Standard Bruce protocol will be used to measure (VO2) max. The Bruce protocol for multi stage treadmill testing of maximal exercise will be used. This will begin with stage 1 with walking slowly for three minutes at 2.7 Km/hr at a 10% grade (inclination), speed and grade then increased in every stage of 3 minutes and end at stage 7 or till exhaustion.
Assessing the change in body weight | Baseline and 2 months post-intervention
  Assessment via using of body weight scale with height (m) scale to be able to calculate body weight (Kg).
Assessing the change in waist hip circumference | Baseline and 2 months post-intervention
  Assessment via using Tape measures It will be used to measure waist and hip circumference and calculate waist hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Manar Elbaz, Demonstrator, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No